CLINICAL TRIAL: NCT05745025
Title: Repeated Transcranial Magnetic Stimulation and Rehabilitation for Individuals With Complex Regional Pain Syndrome Type 1
Brief Title: rTMS and Rehabilitation for Individuals With CRPS Type 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Reflex Sympathetic Dystrophy Syndrome Association (RSDSA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1809306-4
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Complex Regional Pain Syndrome Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, providers of physical therapy, primary investigator, and outcome assessor will be blinded to group allocation. The provider delivering the rTMS will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS and Rehabilitation (Experimental): Subjects in this arm will get rTMS to the contralateral motor cortex and best practice rehabilitation.
  Interventions: Device: Repeated Transcranial Magnetic Stimulation; Other: Rehabilitation
- Sham rTMS and Rehabilitation (Sham Comparator): Subjects in this arm will get sham rTMS to the contralateral motor cortex and best practice rehabilitation.
  Interventions: Device: Sham Repeated Transcranial Magnetic Stimulation; Other: Rehabilitation

INTERVENTIONS:
Device: Repeated Transcranial Magnetic Stimulation — rTMS will be delivered using a commercially available magnetic stimulator (Rapid2, Magstim Inc., Eden Prairie, MN) with a figure-of-8 Air Film coil at 10 Hz. Coil orientation will be optimized for stimulation of the abductor pollicis brevis. Stimulation targeting will be identified using motor-evoked potentials (MEP) of the first dorsal interossei that will be monitored using electromyography (EMG) (Motion Lab Systems Inc., Baton Rouge, LA). The motor threshold (MT) of the muscle will then be identified by systematically adjusting the pulse intensity. The MT will be considered the lowest stimulation intensity at which 5 out of 10 MEPs have a peak-to-peak amplitude of at least 50 microvolts. rTMS will be performed at the identified optimal location at 10Hz using an intensity that is 80% of the MT. Pulse trains will be delivered for 10 seconds, with a 30-second rest for 20 repetitions.
  Other Names: rTMS
  Arms: rTMS and Rehabilitation
Device: Sham Repeated Transcranial Magnetic Stimulation — Sham rTMS will be performed using the same methods as the active group, but a sham Air Film coil (Magstim Inc., Eden Prairie, MN) will be used. This coil looks and sounds like the active coil, but it does not deliver magnetic pulses.
  Other Names: SrTMS
  Arms: Sham rTMS and Rehabilitation
Other: Rehabilitation — Rehabilitation will consist of education, value-based goal setting, Graded Motor Imagery (GMI) (3 components described below), and graded activity. Subjects will complete activities at treatment sessions and be asked to perform certain treatment activities at home.
  Week 1: Pain education, functional value-based goal setting, laterality training (first component of GMI), one task for graded activity (task-based on patient goals)
  Week 2: Continue week 1 activity, add graded motor imagery (second component of GMI), progress 1st graded activity, and initiate 2nd graded activity exercise.
  Week 3- Mirror therapy (third component of GMI), assess knowledge and update education as needed, progress graded activity 1 and 2, and add 3rd graded activity if appropriate based on patient goals.
  Week 4- Continue with week 3 activities. Discuss experience with meditation and progress graded activity as tolerated

SUMMARY:
Subjects with complex regional pain syndrome (CRPS) Type 1 will be randomized to receive repeated transcranial magnetic stimulation (rTMS) followed by rehabilitation or sham rTMS followed by rehabilitation. Treatment will last for 4 weeks, with the first week including 4 rTMS treatments and 2 rehabilitation treatments. Subsequent weeks will include 2 rTMS treatments followed by 2 rehabilitation treatments. Outcome measures will include pain ratings, PROMIS questionnaires, global rating of change, and grip strength or 1 repetition maximum leg press.

DETAILED DESCRIPTION:
Subjects will be randomized to receive either real or sham rTMS, combined with rehabilitation. Subjects will attend 10 sessions over 4 weeks.

rTMS will be delivered at 10Hz using an intensity of 80% of the motor threshold. Pulse trains will be delivered for 10 seconds, with a 30-second rest for 20 repetitions. This will result in a total of 2,000 pulses of magnetic stimulation and will take approximately 20 minutes. There will be 10 rTMS sessions over the 4 weeks.

Sham rTMS will be delivered using the same method as rTMS, but a sham coil, that does not deliver magnetic stimulation, will be used.

Rehabilitation will include graded motor imagery, education, and graded functional activity. There will be 8 rehabilitation sessions over 4 weeks.

Outcomes will include questionnaires asking about pain and function, and either grip strength or leg press strength measurements.

ELIGIBILITY:
Inclusion Criteria:

* Upper or lower extremity CRPS Type 1 (also called RSD-Reflex Sympathetic Dystrophy) of at least 6 months.
* Pain rating on NPRS of at least 4/10
* No initiation of a new intervention (i.e., medication, rehab, injections) in the previous 2 months.
* No plan to initiate a new intervention during the study treatment timeframe (4 weeks).

Exclusion Criteria:

* A history of seizures or epilepsy
* Intracranial metallic devices
* Pacemaker
* Intrathecal infusion pumps
* Brain or spinal cord stimulators with epidural electrodes
* Other ferromagnetic metallic intracranial implants
* Apparent mental or psychiatric disorder that prevents adequate informed consent
* Current pregnancy
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) Weekly Average | Sessions 1 (week 1), 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4). Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session.
  Subjects will be asked to rate their weekly average pain on a scale from 0-10 (0 indicating no pain and 10 indicating worse possible pain).

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) worse/least pain over 24 hours | Sessions 1 (week 1), 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4). Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session
  Subjects will be asked to rate their highest pain level and lowest pain level over a 24-hour period. (0 indicating no pain and 10 indicating worse possible pain).
Patient-Reported Outcomes Measurement Information Systems (PROMIS). | Sessions 1 (week 1), 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4). Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session
  NIH developed computer adaptive tools measuring pain interference, pain behavior, physical functioning, social roles, fatigue, depression, anxiety, and anger. Scores are reported based on T-scores with a mean population score of 50 and a standard deviation of 10. Scores generally range from 20-80. For symptom scales (i.e. pain interference), higher scores indicate worse symptoms, and for function scales (i.e. social roles), higher scores indicate better function.
Global Rating of Change (GROC) | Sessions 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4). Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session
  Subjects will be asked to rate the change of their symptoms from 7(a great deal better) to -7 (a great deal worse) with 0 being no different.
Global Rating of Change Impact (GROCi) | Sessions 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4) Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session
  Subjects will be asked to rate the impact of the change from 7(a great deal better) to -7 (a great deal worse) with 0 being no different.
Patient Acceptable Symptom State (PASS) | Sessions 1 (week 1), 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4). Surveys will also be sent at 4 weeks, 3 months, 6 months, and 1 year after last session.
  Patients are asked if their current state of symptoms is acceptable, yes/no
Grip Strength or 1 Rep Leg Press | Sessions 1 (week 1), 4 (week 1), 6 (week 2), 8 (week 3), 10 (week 4).
  Subjects with upper extremity involvement will have grip strength measured using a dynamometer. Subjects with lower extremity involvement will be tested with single leg 1 rep max leg press.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rufa, DPT, PhD, Principal Investigator — SUNY Upstate Medical Univerity
Locations (1):
- SUNY Upstate Medical Univeristy Institute of Human Performance, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shafiee E, MacDermid J, Packham T, Walton D, Grewal R, Farzad M. The Effectiveness of Rehabilitation Interventions on Pain and Disability for Complex Regional Pain Syndrome: A Systematic Review and Meta-analysis. Clin J Pain. 2023 Feb 1;39(2):91-105. doi: 10.1097/AJP.0000000000001089. PMID 36650605
- [Background] Eldufani J, Elahmer N, Blaise G. A medical mystery of complex regional pain syndrome. Heliyon. 2020 Feb 19;6(2):e03329. doi: 10.1016/j.heliyon.2020.e03329. eCollection 2020 Feb. PMID 32149194
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Picarelli H, Teixeira MJ, de Andrade DC, Myczkowski ML, Luvisotto TB, Yeng LT, Fonoff ET, Pridmore S, Marcolin MA. Repetitive transcranial magnetic stimulation is efficacious as an add-on to pharmacological therapy in complex regional pain syndrome (CRPS) type I. J Pain. 2010 Nov;11(11):1203-10. doi: 10.1016/j.jpain.2010.02.006. Epub 2010 Apr 28. PMID 20430702
- [Background] Gaertner M, Kong JT, Scherrer KH, Foote A, Mackey S, Johnson KA. Advancing Transcranial Magnetic Stimulation Methods for Complex Regional Pain Syndrome: An Open-Label Study of Paired Theta Burst and High-Frequency Stimulation. Neuromodulation. 2018 Jun;21(4):409-416. doi: 10.1111/ner.12760. Epub 2018 Mar 4. PMID 29504190
- [Background] Pleger B, Janssen F, Schwenkreis P, Volker B, Maier C, Tegenthoff M. Repetitive transcranial magnetic stimulation of the motor cortex attenuates pain perception in complex regional pain syndrome type I. Neurosci Lett. 2004 Feb 12;356(2):87-90. doi: 10.1016/j.neulet.2003.11.037. PMID 14746870

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT05745025/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT05745025/ICF_001.pdf